CLINICAL TRIAL: NCT02949297
Title: Expanding Patient Applicability With Polymer Sealing Ovation Alto Stent Graft Investigational Device Exemption (IDE) Study
Acronym: ELEVATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Endologix (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 771-0013
Record Dates: First submitted 2016-10-21; First posted 2016-10-31 (Estimated); Results first posted 2021-12-22 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-11

CONDITIONS: Aortic Aneurysm, Abdominal
Keywords: abdominal; aortic; aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Ovation Alto Abdominal Stent Graft System (Other): Endovascular repair of AAA using the Ovation Alto Abdominal Stent Graft System.
  Interventions: Device: Ovation Alto Abdominal Stent Graft System

INTERVENTIONS:
Device: Ovation Alto Abdominal Stent Graft System — Repair of Abdominal Aortic Aneurysm with Ovation Alto Abdominal Stent Graft System

SUMMARY:
A prospective clinical evaluation of the effectiveness of the Ovation Alto Abdominal Stent Graft System when used in the treatment of subjects with abdominal aortic aneurysm (AAA).

DETAILED DESCRIPTION:
A prospective clinical evaluation of the effectiveness of the Ovation Alto Abdominal Stent Graft System when used in the treatment of subjects with abdominal aortic aneurysm (AAA). The primary objective is to evaluate treatment success at 12 months with the Ovation Alto Abdominal Stent Graft system. The study will have up to 16 sites, and up to 75 patients based on attrition rates. The follow-up intervals will be at 1, 6, and 12 months following initial implant procedure.

ELIGIBILITY:
Inclusion Criteria include:

1. Patient has adequate iliac/femoral access compatible with the required delivery systems.
2. Patient has non-aneurysmal proximal aortic neck.
3. Patient has non-aneurysmal distal iliac landing zone.

Exclusion Criteria include:

1. Patient has dissecting aneurysm.
2. Patient has acutely ruptured aneurysm.
3. Patient has need for emergent surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2017-03-30 (Actual); Primary Completion 2019-03-06 (Actual); Study Completion 2019-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sean Lyden, MD, Principal Investigator — The Cleveland Clinic
Locations (13):
- United States (13):
  - Abrazo Arizona Heart Hospital, Phoenix, Arizona
  - VA San Diego, San Diego, California
  - Northwestern University, Chicago, Illinois
  - Carle Foundation Hospital, Urbana, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - New Mexico Heart Institute, Albuquerque, New Mexico
  - University at Buffalo Clinical Translational Research Center/Kaleida Health/GVI/Buffalo General Medical Center, Buffalo, New York
  - Mission Hospital, Asheville, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - North Central Heart, Sioux Falls, South Dakota
  - Wellmont CVA Heart Institute, Kingsport, Tennessee
  - Baylor St. Luke's Medical Center, Houston, Texas
  - Swedish Heart and Vascular Research, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lyden SP, Metzger DC, Henao S, Noor S, Barleben A, Henretta JP, Kirksey L. One-year safety and effectiveness of the Alto abdominal stent graft in the ELEVATE IDE trial. J Vasc Surg. 2023 Feb;77(2):446-453.e3. doi: 10.1016/j.jvs.2022.08.016. Epub 2022 Aug 24. PMID 36028158
- See also: Endologix Website — http://www.endologix.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Ovation Alto Abdominal Stent Graft System: Endovascular repair of abdominal aortic aneurysm (AAA) using the Ovation Alto Abdominal Stent Graft System.
  Ovation Alto Abdominal Stent Graft System: Repair of Abdominal Aortic Aneurysm with Ovation Alto Abdominal Stent Graft System
Period: 1 Month
Arm/Group | Ovation Alto Abdominal Stent Graft System
Started | 75
Completed | 75
Not Completed | 0
Period: 6 Months
Arm/Group | Ovation Alto Abdominal Stent Graft System
Started | 75
Completed | 72
Not Completed | 3
Period: 12 Months
Arm/Group | Ovation Alto Abdominal Stent Graft System
Started | 72
Completed | 67
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | Ovation Alto Abdominal Stent Graft System
Number analyzed (Participants) | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 73 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 70
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/not Hispanic or Latino | 58
  White/Hispanic or Latino | 1
  Black or African American/not Hispanic or Latino | 1
  Unknown/not Hispanic or Latino | 11
  Unknown/Hispanic or Latino | 1
  Unknown/Unknown | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 75
Left Ankle Brachial Index [Mean (Standard Deviation); unit: ratio] — The Ankle Brachial Index is the systolic pressure at the ankle, divided by the systolic pressure at the arm. Population: Data point only provided for 73 out of 75 subjects. Reason is unknown why this information was not provided for 2 out of 75 subjects
  ratio
    number analyzed (Participants) | 73
    (all) | 1 (0)
Right Ankle Brachial Index [Mean (Standard Deviation); unit: ratio] — The Ankle Brachial Index is the systolic pressure at the ankle, divided by the systolic pressure at the arm Population: Data point only provided for 72 out of 75 subjects. Reason is unknown why this information was not provided for 3 out of 75 subjects
  ratio
    number analyzed (Participants) | 72
    (all) | 1 (0)
ASA Class [Count of Participants; unit: Participants] — The American Society of Anesthesiologists (ASA) presents a graded scale assessing a subject's risk of undergoing anesthesia. ASA I: A normal healthy patient without any systemic disease, undergoing elective surgery ASA II: A patient with mild systemic disease. Disease does not affect daily activities.
  ASA III: Individual with multiple system disease or well controlled major system disease. Disease does limit daily activities.
  ASA IV: Individual in imminent danger of death. Surgery is viewed to be last resort at salvaging life. Individual not expected to live through the next 24 hours.
  Participants
    Class 1/2 | 5
    Class 3/4 | 70
Height [Mean (Standard Deviation); unit: cm] | 179 (9)
Weight [Mean (Standard Deviation); unit: kilograms] | 95 (19)
Calculated BMI [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index (BMI) is a person's weight in kilograms divided by the square of height in meters
  kg/m^2 | 30 (5)
Cardiovascular History [Count of Participants; unit: Participants]
  Coronary Artery Disease | 35
  Prior PTCA | 3
  Prior CABG | 5
  Stents | 7
  Valvular Heart Disease | 11
  Prior Valve Repair | 0
  Prior Valve Replacement | 2
  Angina pectoris or chest discomfort | 5
  Cardiomyopathy | 3
  Congestive Heart Failure | 6
  Myocardial Infarction | 11
  Arrhythmia | 17
  Pacemaker | 3
  ICD | 1
  AICD | 0
  Anticoagulant medication | 7
  Hypertension | 62
  Hypotension | 0
  Hyperlipidemia | 57
  Other | 10
Peripheral Vascular, Stroke, and Aneurysm History [Count of Participants; unit: Participants]
  Peripheral Vascular Disease | 13
  Atherosclerosis | 8
  Thromboangiitis obliterans | 0
  Chronic Venous Insufficiency | 2
  Claudication | 4
  Deep Venous Thrombosis | 3
  Peripheral Embolism | 2
  Raynauds Phenomenon | 0
  Thrombophlebitis | 0
  Varicose Veins | 1
  Prior surgical repair | 0
  Prior stent | 0
  Carotid artery disease | 6
  Prior carotid artery stenting | 0
  Prior carotid endarterectomy | 1
  Transient Ischemic attacks | 4
  Stroke | 0
  Aneurysms | 75
  Abdominal Aortic Aneurysm | 75
  Cerebral Aneurysm | 0
  Thoracic Aortic Aneurysm | 1
  Family History of Aneurysms | 9
  Other | 8
Pulmonary History [Count of Participants; unit: Participants]
  COPD | 27
  Asthma | 5
  Pneumonia | 4
  Pulmonary Edema | 0
  Pulmonary Embolism | 4
  Respiratory depression or failure | 0
  Mechanical ventilation >24 hours | 0
  Obstructive sleep apnea | 14
  Tobacco Use (Current) | 15
  Tobacco Use (former) | 56
  Other | 16
Gastrointestinal, Genitourinary, Reproductive History [Count of Participants; unit: Participants]
  Renal Insufficiency | 5
  Receiving any form of dialysis | 0
  Chronic Renal Failure | 0
  Renal Microemboli | 0
  Chronic urinary tract infections | 1
  Incontinence bladder problems | 3
  Gastrointestinal bleeding | 2
  Bowel ischemia | 0
  Bowel obstruction | 1
  Bowel fistulas | 0
  Paralytic or adynamic ileus | 0
  Impotence including erectile dysfunction | 8
  Other | 42
Neurological History [Count of Participants; unit: Participants]
  Reversible Ischemic Neurologic Disease | 0
  Paraplegia | 0
  Parasthesia | 1
  Chronic Back Pain | 18
  Chronic Headaches, Migraines | 3
  Other | 20
Endocrine History [Count of Participants; unit: Participants]
  Diabetes Type I | 0
  Diabetes Type II | 22
  Diabetic incompressible vessels | 0
  Immunodeficiency | 2
  Hyperthyroidism or Hypothyroidism | 8
  Other | 5
Hematological History [Count of Participants; unit: Participants]
  Hemorrhage | 0
  Coagulopathy disorder | 0
  Anemia | 5
  Platelet Disorder | 0
  Other | 5
Psychosocial History [Count of Participants; unit: Participants]
  Depression | 7
  Prior substance abuse | 1
  Alcohol | 3
  Illicit drugs | 0
  Other | 4
Miscellaneous Medical History [Count of Participants; unit: Participants]
  Connective Tissue Disorder | 0
  Allergy, Intolerance to PTFE, polymers, FEP, nitinol | 0
  Hypersensitivity to anticoagulation, contrast | 0
  Cancer | 14
  Liver Disease | 5
  Other significant medical, surgical history | 26
Juxtarenal angle [Mean (Standard Deviation); unit: degrees] | 23.1 (18.7)
Aortic diameter Inferior Renal -35mm [Mean (Standard Deviation); unit: mm]
  Minimum | 25.0 (2.3)
  Maximum | 26.6 (2.4)
  Average | 25.9 (2.3)
Aortic diameter inferior renal [Mean (Standard Deviation); unit: mm]
  Minimum | 21.8 (2.5)
  Maximum | 23.2 (2.6)
  Average | 22.5 (2.5)
Aortic diameter inferior renal +7mm [Mean (Standard Deviation); unit: mm]
  Minimum | 21.8 (2.3)
  Maximum | 23.0 (2.7)
  Average | 22.4 (2.4)
Change from diameter at inferior renal artery to inferior renal artery diameter at +7mm [Mean (Standard Deviation); unit: %] — This is the percentage of change from the diameter at the lowest inferior renal artery to the diameter at inferior renal artery +7mm.
  % | 0.0 (7.2)
Aortic diameter inferior renal +10mm [Mean (Standard Deviation); unit: mm]
  Minimum | 21.8 (2.5)
  Maximum | 23.4 (2.8)
  Average | 22.6 (2.5)
Maximum Sac Diameter [Count of Participants; unit: Participants]
  <40 mm | 4
  ≥40, <50 mm | 23
  ≥ 50, <60 mm | 40
  ≥ 60 mm | 8
Native Bifurcation [Mean (Standard Deviation); unit: mm] — Population: Data point only provided for 74 of 75 subjects.
  mm
    Minimum: number analyzed (Participants) | 74
    Minimum | 20.1 (5.1)
    Maximum: number analyzed (Participants) | 74
    Maximum | 26.2 (6.7)
Transverse dimension of adjacent normal aortic segment [Mean (Standard Deviation); unit: mm] | 22.7 (4.1)
Neck Length [Mean (Standard Deviation); unit: mm] | 27.9 (13.7)
Distance from the most distal renal artery to most superior left internal iliac artery [Mean (Standard Deviation); unit: mm] | 182.5 (24.7)
Distance from the most distal renal artery to most superior right internal iliac artery (mm) 75 181. [Mean (Standard Deviation); unit: mm] | 181.2 (21.0)
Inferior Renal to Aortic Bifurcation [Mean (Standard Deviation); unit: mm] | 110.9 (13.1)
Right Distal Iliac Diameter [Mean (Standard Deviation); unit: mm]
  Minimum | 15.8 (3.8)
  Maximum | 17.1 (4.0)
  Average | 16.5 (3.9)
Right external iliac diameter [Mean (Standard Deviation); unit: mm]
  Minimum | 7.6 (1.6)
  Maximum | 8.7 (1.6)
  Average | 8.1 (1.5)
Left distal iliac diameter [Mean (Standard Deviation); unit: mm]
  Minimum | 15.1 (3.0)
  Maximum | 16.4 (3.3)
  Average | 15.8 (3.1)
Left external iliac diameter [Mean (Standard Deviation); unit: mm]
  Minimum | 7.6 (1.9)
  Maximum | 8.7 (1.6)
  Average | 8.2 (1.7)
Left distal iliac landing zone [Mean (Standard Deviation); unit: mm] | 49.1 (18.7)
Right distal iliac landing zone [Mean (Standard Deviation); unit: mm] | 50.1 (20.7)
SIR Calcification Grade [Count of Participants; unit: Participants] — Amount of calcium present in the cross-sectional area of the target location of the sealing ring
  Participants
    Calcification 0% of circumference | 14
    Calcification <25% of circumference | 49
    Calcification 25-50% of circumference | 11
    Calcification >50% of circumference | 1
SIR Thrombus Grade [Count of Participants; unit: Participants] — Amount of thrombus present in the cross-sectional area of the target location of the sealing ring
  Participants
    Thrombus 0% of circumference | 27
    Thrombus <25% of circumference | 16
    Thrombus 25-50% of circumference | 18
    Thrombus >50% of circumference | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Treatment Success
Description: Treatment success is defined as technical success, freedom from type I and III endoleaks at 12 months, freedom from stent graft migration > 10m at 12 months compared to 1 month baseline, freedom from AAA enlargement >5mm at 12 months (compared to 1-month baseline, freedom from AAA rupture through 12 months, freedom from conversion to open repair through 12 months, stent graft stenosis, occlusion or kink requiring secondary intervention through 12 months, thromboembolic event attributable to stent graft requiring secondary intervention through 12 months, stent fracture requiring secondary intervention through 12 months.
Time Frame: 12 months
Population: 61 subjects were evaluable at 1 year- evaluable meaning able to be assessed for all items of composite endpoint of treatment success; 67 subjects completed 1 year, however, some of these subjects did not have imaging or imaging was not evaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Ovation Alto Abdominal Stent Graft System
Number analyzed (Participants) | 61
Participants | 58
Statistical Analysis 1: Comparison: Ovation Alto Abdominal Stent Graft System; Test type: Other — One-sided Clopper-Pearson 95% confidence interval; Clopper-Pearson = 80, 95% CI 1-sided [upper limit 95] — One-sided Clopper-Pearson 95% confidence interval

2. Secondary Outcome: Event Rates for Endoleaks
Description: Endoleak is defined by the persistence of blood flow outside the lumen of the endovascular graft but within the aneurysm sac and can be classified as:
  * Type I - Ineffective seal at either the proximal or distal sealing zones
    * Type IA - Ineffective seal at the proximal sealing zone
    * Type IB - Ineffective seal at the distal sealing zone
  * Type II - Retrograde blood flow from lumbar arteries, the inferior mesenteric artery, or other collateral vessels into the aneurysm sac
  * Type III - A leak caused by fabric tears or disruption, component disconnection, or graft disintegration
  * Type IIIA - Junctional leak or component disconnection
  * Type IIIB - Midgraft hole
  * Type IV - Blood flow through an intact fabric.
  * Unknown endoleak - Endoleak present but unable to assess type Endoleak will only be evaluated as an adverse event or serious adverse event if it is present at the 30-day follow-up visit or if a post-index procedure re-intervention occurs.
Time Frame: 1 month, 6 months, 12 months
Population: All available data has been analyzed; due to imagining requirements and quality of imaging, all patients present for visit may not have been evaluable per definitions.
Measure: Number; unit: endoleaks
Arm/Group | Ovation Alto Abdominal Stent Graft System
Number analyzed (Participants) | 75
endoleaks
  1 month : Type I: number analyzed (Participants) | 73
  1 month : Type I | 0
  1 month : Type Ia: number analyzed (Participants) | 73
  1 month : Type Ia | 1
  1 month : Type Ib: number analyzed (Participants) | 73
  1 month : Type Ib | 0
  1 month : Type II: number analyzed (Participants) | 73
  1 month : Type II | 34
  1 month : Type III: number analyzed (Participants) | 73
  1 month : Type III | 0
  1 month : Type IIIA: number analyzed (Participants) | 73
  1 month : Type IIIA | 0
  1 month : Type IIIB: number analyzed (Participants) | 73
  1 month : Type IIIB | 0
  1 month : Type IV: number analyzed (Participants) | 73
  1 month : Type IV | 0
  1 month : Unknown: number analyzed (Participants) | 73
  1 month : Unknown | 3
  6 month : Type I: number analyzed (Participants) | 70
  6 month : Type I | 0
  6 month : Type Ia: number analyzed (Participants) | 70
  6 month : Type Ia | 0
  6 month : Type Ib: number analyzed (Participants) | 70
  6 month : Type Ib | 0
  6 month : Type II: number analyzed (Participants) | 70
  6 month : Type II | 30
  6 month : Type III: number analyzed (Participants) | 70
  6 month : Type III | 0
  6 month : Type IIIA: number analyzed (Participants) | 70
  6 month : Type IIIA | 0
  6 month : Type IIIB: number analyzed (Participants) | 70
  6 month : Type IIIB | 0
  6 month : Type IV: number analyzed (Participants) | 70
  6 month : Type IV | 0
  6 month : Unknown: number analyzed (Participants) | 70
  6 month : Unknown | 0
  1 year : Type I: number analyzed (Participants) | 61
  1 year : Type I | 0
  1 year : Type Ia: number analyzed (Participants) | 61
  1 year : Type Ia | 0
  1 year : Type Ib: number analyzed (Participants) | 61
  1 year : Type Ib | 0
  1 year : Type II: number analyzed (Participants) | 61
  1 year : Type II | 25
  1 year : Type III: number analyzed (Participants) | 61
  1 year : Type III | 0
  1 year : Type IIIA: number analyzed (Participants) | 61
  1 year : Type IIIA | 0
  1 year : Type IIIB: number analyzed (Participants) | 61
  1 year : Type IIIB | 0
  1 year : Type IV: number analyzed (Participants) | 61
  1 year : Type IV | 0
  1 year : Unknown: number analyzed (Participants) | 61
  1 year : Unknown | 2

3. Secondary Outcome: Number of Participants With Stent Graft Migration > 10mm
Description: any change of stent graft migration (movement) greater than 10mm
Time Frame: 6 months, 12 months
Population: Analysis based on all data available; imaging not available for all subjects to determine migration.
Measure: Count of Participants; unit: Participants
Arm/Group | Ovation Alto Abdominal Stent Graft System
Number analyzed (Participants) | 71
Participants
  6 Months | 0
  1 Year: number analyzed (Participants) | 64
  1 Year | 0

4. Secondary Outcome: Number of Participants With AAA Enlargement > 5mm
Description: Change in aneurysm diameter greater than 5mm
Time Frame: 6 months, 12 months
Population: Subjects lost to follow-up withdrawn, death, or imaging not available.
Measure: Count of Participants; unit: Participants
Arm/Group | Ovation Alto Abdominal Stent Graft System
Number analyzed (Participants) | 72
Participants
  6 months | 0
  12 months: number analyzed (Participants) | 64
  12 months | 1

5. Secondary Outcome: Number of Participants With AAA Rupture
Description: A tear in the abdominal aorta that can result in serious internal bleeding.
Time Frame: 30 day, Day 31-365
Measure: Count of Participants; unit: Participants
Arm/Group | Ovation Alto Abdominal Stent Graft System
Number analyzed (Participants) | 75
Participants
  1 month | 0
  Day 31-365 | 0

6. Secondary Outcome: Number of Participants With Conversion to Open Repair
Description: conversion to open abdominal surgery to repair AAA
Time Frame: 30 day, Day 31-365
Measure: Count of Participants; unit: Participants
Arm/Group | Ovation Alto Abdominal Stent Graft System
Number analyzed (Participants) | 75
Participants
  30 day | 0
  Day 31 to 365 | 1

7. Secondary Outcome: Number of Secondary Interventions
Description: Intervention occurring after index procedure and having to do with device or AAA.
Time Frame: 30 days, Day 31-365
Measure: Count of Participants; unit: Participants
Arm/Group | Ovation Alto Abdominal Stent Graft System
Number analyzed (Participants) | 75
Participants
  1 month | 0
  Day 31 - 365 | 2

8. Secondary Outcome: Number of Participants With AAA-related Mortality
Description: death caused by or related to AAA
Time Frame: 1 month, Day 31-365
Measure: Count of Participants; unit: Participants
Arm/Group | Ovation Alto Abdominal Stent Graft System
Number analyzed (Participants) | 75
Participants
  30 days | 0
  Day 31 to 365 | 0

9. Secondary Outcome: Device-related Adverse Events (AEs)
Description: Device-Related: Event is caused or contributed by any component of the device during delivery, deployment or while the device is in situ post-operatively
Time Frame: 30 days, Day 31-365
Measure: Count of Participants; unit: Participants
Arm/Group | Ovation Alto Abdominal Stent Graft System
Number analyzed (Participants) | 75
Participants
  30 days : Infections and Infestations | 0
  30 days : Product Issues | 1
  Day 31-365 : Infections and Infestations | 1
  Day 31-365 : Product Issues | 0

10. Secondary Outcome: Major Adverse Events
Description: Major adverse events (MAE) are defined as any one of the following events:
  * Death
  * Myocardial Infarction
  * Stroke (excludes TIA)
  * Renal Failure (excludes renal insufficiency)
  * Respiratory Failure (excludes chronic obstructive pulmonary disease (COPD) or pulmonary complications)
  * Paralysis (excludes paraparesis)
  * Bowel Ischemia
  * Procedural Blood Loss (≥1,000 cc)
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Ovation Alto Abdominal Stent Graft System
Number analyzed (Participants) | 75
Participants
  Deaths : 30 days | 0
  Deaths : 31-365 days | 3
  Bowel Ischemia : 30 days | 3
  Bowel Ischemia : 31-365 days | 0
  Myocardial Infarction : 30 days | 0
  Myocardial Infarction : 31-365 days | 1
  Paralysis : 30 days | 0
  Paralysis : 31-365 days | 0
  Renal Failure : 30 days | 0
  Renal Failure : 31-365 days | 0
  Respiratory Failure : 30 days | 0
  Respiratory Failure : 31-365 days | 0
  Stroke : 30 days | 0
  Stroke : 31-365 days | 0
  Procedural Blood Loss >1000cc : 30 days | 1
  Procedural Blood Loss >1000cc : 31-365 days | 0

11. Secondary Outcome: Number of Participants With Other Stent Graft Finding (Includes Kinking and Stent Compression)
Description: The integrity of the stent graft is evaluated by the Independent Core Lab via abdominal X-rays at regularly scheduled follow-up visits. Any fractured stents, and any other issues compromising the integrity of the stent graft will be reported.
Time Frame: 1 month, 6 months, 12 months
Population: Imaging not available for every subject at every timepoint
Measure: Count of Participants; unit: Participants
Arm/Group | Ovation Alto Abdominal Stent Graft System
Number analyzed (Participants) | 74
Participants
  1 Month | 0
  6 Months: number analyzed (Participants) | 72
  6 Months | 0
  1 Year: number analyzed (Participants) | 64
  1 Year | 0

12. Secondary Outcome: Number of Participants With Stent Fracture
Description: as for outcome 11
Time Frame: 1 month, 6 months, 12 months
Population: Subjects lost to follow-up withdrawn, death, or imaging not available.
Measure: Count of Participants; unit: Participants
Arm/Group | Ovation Alto Abdominal Stent Graft System
Number analyzed (Participants) | 70
Participants
  1 month | 0
  6 months: number analyzed (Participants) | 69
  6 months | 0
  12 months: number analyzed (Participants) | 61
  12 months | 0

13. Secondary Outcome: Adverse Events (Serious and Non-serious)
Description: An adverse event is any new, undesirable medical occurrence or change (worsening) of a pre-existing condition that occurs in a subject, whether or not considered to be associated with the product
Time Frame: 30 days, Day 31-365
Measure: Count of Participants; unit: Participants
Arm/Group | Ovation Alto Abdominal Stent Graft System
Number analyzed (Participants) | 75
Participants
  30 days : Blood and lymphatic System Disorder | 0
  30 days : Cardiac Disorder | 0
  30 days : Ear and Labyrinth Disorders | 0
  30 days : Gastrointestinal Disorders | 4
  30 days : General Disorders and Administration Site Conditions | 13
  30 days : Hepatobiliary Disorders | 0
  30 days : Immune System Disorder | 2
  30 days : Infections and Infestations | 5
  30 days : Injury, Poisoning and Procedural Complications | 5
  30 days : Musculoskeletal and Connective Tissue Disorders | 1
  30 days : Neoplasms Benign, Malignant and Unspecified (incl. Cysts and Polyps) | 0
  30 days : Nervous System Disorders | 1
  30 days : Other | 2
  30 days : Product Issues | 1
  30 days : Psychiatric Disorders | 1
  30 days : Renal and Urinary Disorders | 4
  30 days : Respiratory, Thoracic and Mediastinal Disorders | 2
  30 days : Vascular Disorders | 7
  Day 31-365 : Blood and lymphatic System Disorder | 2
  Day 31-365 : Cardiac Disorder | 11
  Day 31-365 : Ear and Labyrinth Disorders | 1
  Day 31-365 : Gastrointestinal Disorders | 3
  Day 31-365 : General Disorders and Administration Site Conditions | 15
  Day 31-365 : Hepatobiliary Disorders | 2
  Day 31-365 : Immune System Disorder | 1
  Day 31-365 : Infections and Infestations | 2
  Day 31-365 : Injury, Poisoning and Procedural Complications | 2
  Day 31-365 : Musculoskeletal and Connective Tissue Disorders | 7
  Day 31-365 : Neoplasms Benign, Malignant and Unspecified (incl. Cysts and Polyps) | 4
  Day 31-365 : Nervous System Disorders | 3
  Day 31-365 : Other | 2
  Day 31-365 : Product Issues | 0
  Day 31-365 : Psychiatric Disorders | 0
  Day 31-365 : Renal and Urinary Disorders | 4
  Day 31-365 : Respiratory, Thoracic and Mediastinal Disorders | 3
  Day 31-365 : Vascular Disorders | 9

14. Secondary Outcome: Procedure-related Adverse Event
Description: Procedure-Related event is caused or contributed by the initial study device implantation (index) procedure, up to 30 days, unless a different etiology can be identified
Time Frame: 30 days, Day 31-365
Measure: Count of Participants; unit: Participants
Arm/Group | Ovation Alto Abdominal Stent Graft System
Number analyzed (Participants) | 75
Participants
  30 days : Gastrointestinal Disorders | 2
  30 days : General Disorders and Administration Site Conditions | 0
  30 days : Injury Poisoning and Procedural Complications | 3
  30 days : Product Issues | 1
  30 days : Vascular Disorders | 0
  Day 31-365 : Gastrointestinal Disorders | 0
  Day 31-365 : General Disorders and Administration Site Conditions | 2
  Day 31-365 : Injury Poisoning and Procedural Complications | 0
  Day 31-365 : Product Issues | 0
  Day 31-365 : Vascular Disorders | 1

15. Secondary Outcome: Serious Adverse Event
Description: A serious adverse event (SAE) defined as one that suggests a significant hazard or side effect, regardless of the investigator or Sponsor's opinion on the relationship to the investigational product. This includes, but may not be limited to, any event that:
  * Is fatal
  * Is life-threatening
  * Requires or prolongs (>48 hours) inpatient hospitalization
  * Is a persistent or significant disability or incapacity
  * Is considered an important medical event
Time Frame: 30 Days, Day31-365)
Measure: Count of Participants; unit: Participants
Arm/Group | Ovation Alto Abdominal Stent Graft System
Number analyzed (Participants) | 75
Participants
  30 days : Cardiac disorders | 0
  30 days : Gastrointestinal Disorders | 2
  30 days : Infections and Infestations | 0
  30 days : Neoplasms Benign, Malignant and Unspecified (incl. Cysts and Polyps) | 0
  30 days : Nervous System Disorders | 0
  30 days : Product Issues | 1
  30 days : Vascular Disorders | 0
  30 days : Injury, Poisoning and Procedural Complications | 2
  Day 31-365 : Cardiac disorders | 2
  Day 31-365 : Gastrointestinal Disorders | 0
  Day 31-365 : Infections and Infestations | 1
  Day 31-365 : Neoplasms Benign, Malignant and Unspecified (incl. Cysts and Polyps) | 1
  Day 31-365 : Nervous System Disorders | 1
  Day 31-365 : Product Issues | 0
  Day 31-365 : Vascular Disorders | 1
  Day 31-365 : Injury, Poisoning and Procedural Complications | 0

ADVERSE EVENTS:
Time Frame: AEs were collected over 1 year.
Arm/Group | Ovation Alto Abdominal Stent Graft System
All-Cause Mortality (participants affected / at risk) | 3/75
Serious Adverse Events (participants affected / at risk) | 11/75
Other Adverse Events (participants affected / at risk) | 54/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ovation Alto Abdominal Stent Graft System (N=75)
Bowel Ischemia (Gastrointestinal disorders) | 3
Endoleak Ia (Product Issues) | 1
Aneurysm Expansion (Vascular disorders) | 1
Procedural Blood Loss (Injury, poisoning and procedural complications) | 1
Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Device Infection (Infections and infestations) | 1
Other (Nervous system disorders) | 1 — Lewy body dementia contributed to the patient's recurrent falls and ultimately expiration
Myocardial Infarction (Cardiac disorders) | 1
Unknown Cause of Death (Cardiac disorders) | 1 — Efforts to figure out cause of death were unsuccessful x3.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ovation Alto Abdominal Stent Graft System (N=75)
anemia (Blood and lymphatic system disorders) | 2
Acute Renal Failure (Renal and urinary disorders) | 2
Adynamic Ileus (Gastrointestinal disorders) | 1
Angina (Cardiac disorders) | 1
Anticoagulant Related Bleeding (General disorders) | 1
Arrhythmia (Cardiac disorders) | 3
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Bone Fracture (Musculoskeletal and connective tissue disorders) | 1
Claudication (Vascular disorders) | 2
Congestive Heart Failure (Cardiac disorders) | 3
COPD (Infections and infestations) | 1
Deep Vein Thrombosis (Vascular disorders) | 1
Edema (Cardiac disorders) | 1
Embolism (Vascular disorders) | 1
Endoleak IA (General disorders) | 1
Endoleak II (General disorders) | 27
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Medication Reaction (Immune system disorders) | 1
Medication Reaction (General disorders) | 1
Numbness (General disorders) | 1
Routine CT scan done for follow up of AAA stent graft repair (Gastrointestinal disorders) | 1
plaque obstructing true lumen (iliofemoral endarterectomy) (Vascular disorders) | 1
Hematuria (Injury, poisoning and procedural complications) | 1
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1
Blood in urine (Renal and urinary disorders) | 1
hypoxemia (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia (Infections and infestations) | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1
Sub-Dermal Hematoma (Injury, poisoning and procedural complications) | 1
Syncope (Cardiac) (Cardiac disorders) | 1
Syncope (cardiac) (Nervous system disorders) | 1
TIA (Nervous system disorders) | 1
Urinary Retention (Renal and urinary disorders) | 1
UTI (Infections and infestations) | 3
Valve Disorder (Cardiac disorders) | 1
Restrictive lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1
Proglide failure during surgical closure of left groin incision (Vascular disorders) | 1 — Proglide failure during surgical closure of left groin incision
Hematuria (Renal and urinary disorders) | 1
degenerative changes to the body wall (Injury, poisoning and procedural complications) | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1
Ulnar Mononeuropathy (Nervous system disorders) | 1
Bilateral Popliteal Artery Aneurysms (Vascular disorders) | 1
Altered mental status (Nervous system disorders) | 1
Acute Hypoxic Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1
Thoracic Aortic Aneurysm (Vascular disorders) | 1
Choledocholithiasis (Hepatobiliary disorders) | 1
Gout (Immune system disorders) | 1
diarrhea (Gastrointestinal disorders) | 2 — diarrhea
decreased pulse in right foot (Injury, poisoning and procedural complications) | 1
pain in the toes of the right foot (Injury, poisoning and procedural complications) | 1
Pain in right foot with toe discoloration (Musculoskeletal and connective tissue disorders) | 1
MRSA and Enterococcus of the right 4th toe (Infections and infestations) | 1
left plank pain (Infections and infestations) | 1
Severe osteoarthritis right hip (Musculoskeletal and connective tissue disorders) | 1
left testicular infarction (Renal and urinary disorders) | 1
left leg pain (Musculoskeletal and connective tissue disorders) | 1
Nausea (Injury, poisoning and procedural complications) | 1
Post Implant Syndrome (Injury, poisoning and procedural complications) | 1
Acute exacerbation of chronic lower back pain (General disorders) | 1
Polymyalgia Rheumatica (Immune system disorders) | 1
Sciatica pain (Musculoskeletal and connective tissue disorders) | 1
Right forearm bruising (Musculoskeletal and connective tissue disorders) | 1
Encephalopathy (Psychiatric disorders) | 1
Left breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
carotid stenosis (Vascular disorders) | 1
swelling of right leg below the knee (Musculoskeletal and connective tissue disorders) | 1
colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
cholecystectomy (Hepatobiliary disorders) | 1
cataract surgery (Ear and labyrinth disorders) | 1
head laceration (due to fall) (General disorders) | 1
constipation (Gastrointestinal disorders) | 1
right foot pain (General disorders) | 1
benign lung nodule (Respiratory, thoracic and mediastinal disorders) | 1
Hypovolemia (Cardiac disorders) | 1
AKI on CKD (Renal and urinary disorders) | 1
Left ventricular outflow tract obstruction (Cardiac disorders) | 1
Sleeplessness due to PTSD (General disorders) | 1
Prostatitis (Renal and urinary disorders) | 1
Esophageal Stricture (Gastrointestinal disorders) | 1
Hypokalemia (General disorders) | 1
air leak status post left lobectomy (Injury, poisoning and procedural complications) | 1
Endoleak (unknown) (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI can publish institution's data/results 18 months after study conclusion at all sites or when multi-center results are published or notification that results will not be published. Institution is to submit drafts of manuscripts to Endologix 30 days prior to submission for publication or presentation.

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-08-23): https://cdn.clinicaltrials.gov/large-docs/97/NCT02949297/Prot_SAP_ICF_000.pdf